CLINICAL TRIAL: NCT00155961
Title: Odense Androgen Study in the Elderly
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Other Study IDs: 016
Record Dates: First submitted 2005-09-06; First posted 2005-09-12 (Estimated); Last update posted 2006-02-03 (Estimated); Status verified 2005-09

CONDITIONS: Bone Diseases; Metabolic Syndrome
Keywords: Androgens; Metabolic syndrome; Bone mineral density; Body composition; Questionnaire
MeSH Terms: conditions — Bone Diseases; Metabolic Syndrome

STUDY DESIGN:
Time Perspective: Other

SUMMARY:
Introduction

Male ageing is associated with sarcopenia, frailty, osteopenia, obesity, the metabolic syndrome and cardiovascular disease. To what extent the androgens affect these signs of ageing is still largely undetermined. A few studies have shown divergent results concerning the relation between ageing and serum levels of testosterone. It still remains to be shown whether there is a pure age-related decline in serum testosterone or whether other factors such as obesity, chronic illness or medication are responsible for the lower serum testosterone found in elderly men when compared with young men. To investigate these issues a cohort of 600 men aged 60 to 75 years is examined.

Objective

The aim of the study is to investigate the relation of testosterone (T) to body composition (BC) and physical performance (PP). Measures for BC are muscle mass (MM), bone mineral density (BMD) and fat mass (FM). Parameters for PP are maximum voluntary force (MVF), maximum oxygen uptake (VO2max) and muscle power (P). We hypothesize that T is positively associated with MM, BMD and all PP parameters, but negatively associated with FM. We will furthermore examine whether life style, medication, chronic disease, hormones and binding proteins exert their actions on BC and PP solely through or independently of T. The levels of s-total and free T in this cohort will be compared with the s-total and free T levels from a cohort of young men aged 20 to 30 years. Furthermore the associations found between T and BC and PP in the two cohorts will be compared to investigate whether T plays the same role in the two groups.

DETAILED DESCRIPTION:
Introduction

Male ageing is associated with sarcopenia, frailty, osteopenia, obesity, the metabolic syndrome and cardiovascular disease. To what extent the androgens affect these signs of ageing is still largely undetermined. A few studies have shown divergent results concerning the relation between ageing and serum levels of testosterone. It still remains to be shown whether there is a pure age-related decline in serum testosterone or whether other factors such as obesity, chronic illness or medication are responsible for the lower serum testosterone found in elderly men when compared with young men. To investigate these issues a cohort of 600 men aged 60 to 75 years is examined.

Objective

The aim of the study is to investigate the relation of testosterone (T) to body composition (BC) and physical performance (PP). Measures for BC are muscle mass (MM), bone mineral density (BMD) and fat mass (FM). Parameters for PP are maximum voluntary force (MVF), maximum oxygen uptake (VO2max) and muscle power (P). We hypothesize that T is positively associated with MM, BMD and all PP parameters, but negatively associated with FM. We will furthermore examine whether life style, medication, chronic disease, hormones and binding proteins exert their actions on BC and PP solely through or independently of T. The levels of s-total and free T in this cohort will be compared with the s-total and free T levels from a cohort of young men aged 20 to 30 years. Furthermore the associations found between T and BC and PP in the two cohorts will be compared to investigate whether T plays the same role in the two groups.

Methods

All blood analyses are determined in fasting condition from venous samples drawn between 8 and 9 a.m. The influence of life style, medication, chronic disease, hormones and binding proteins on T, BC and PP are assessed by four questionnaires, a physical examination and blood tests. MM is determined regionally (truncal, lower and upper extremities) and as total by Dual Energy X-ray Absorptiometry (DEXA), and specifically by MRI with cross sectional area of femoral and axial muscles. MVF of m. biceps brachii and m. triceps surae is measured isometrically. P is measured with the Nottingham Powerrig. VO2max is determined on a Monark ergometer bike using a Jaeger Oxycon Pro. BMD is determined specifically (femoral and lumbar) as well as total bone mass is estimated by DEXA. The ratio of intraperitoneal area/volume of fat to total abdominal area/volume is determined by MRI, and likewise is also abdominal subcutaneous FM. Finally BMI and waist-to-hip ratio are measured.

Results

Initially a questionnaire providing us with basic demographic, social, occupational and other information about men from Funen aged 60 to 75 was randomly mailed to 4,964 men. Of these questionnaires, 89% were returned and 85.2% of the returned questionnaires had been completed. Afterwards 1,650 people received an invitation by mail to get an introduction to the project via telephone. Of these 1,650 people 50.8% accepted to be contacted. So far 762 people have been contacted in a randomly manner and of these people, 74% have agreed to participate in the project. In the beginning of April 2005, 550 people have been included in Odense Androgen Study in the Elderly.

ELIGIBILITY:
Inclusion Criteria:

* Age: 60-75 years

Exclusion Criteria:

* Cancer
* Severe chronic disease
* Opioid drug addiction

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2002-03

CONTACTS AND LOCATIONS:
Overall Officials: Claus Hagen, MD, DMSc, Principal Investigator — Gentofte County Hospital
Locations (1):
- Department of Endocrinology, Odense University Hospital, Odense, Funen, Denmark

REFERENCES:
- [Derived] Glintborg D, Nielsen TL, Wraae K, Hougaard D, Gudex C, Brixen K, Andersen M. The relationship between health-related quality of life, obesity and testosterone levels in older men. Age Ageing. 2014 Mar;43(2):280-4. doi: 10.1093/ageing/aft203. Epub 2013 Dec 29. PMID 24375324